CLINICAL TRIAL: NCT02118896
Title: A Long-term Follow up Study to Evaluate the Safety and Efficacy in Transplant Recipients Treated With Modified Release Tacrolimus, FK506E (MR4), Based Immunosuppression Regimen
Brief Title: Study to Ascertain if Prolonged Release Tacrolimus (FK506E - MR4) is Safe and Effective When Used in the Long Term and in Combination With Other Immunosuppressive Drugs in Patients Who Have Received a Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F506-CL-0857; 2005-005714-20 (EudraCT Number); FG-506-14-02 (Other: Sponsor Protocol Number)
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplantation; Liver Transplantation; Kidney Transplantation
Keywords: FK506E; Heart Transplantation; MR4; Tacrolimus; Advagraf; Kidney Transplantation; Renal Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: FK506E (MR4) (Experimental): Single open arm of FK506E (MR4). Since this was an extension study for many studies, generally the dose given at enrollment was to be continued. The investigator was permitted to adjust the subject's dose and modify the MR4 dose regimen as deemed necessary to minimize Adverse Events (AEs) and maintain effective immunosuppression. MR4 capsules were taken orally, once daily in the morning. MR4 capsules were to be swallowed with fluid (preferably water) on an empty stomach or at least 1 hour before or 2 to 3 hours after a meal. MR4 was supplied as 0.5 mg, 1 mg and 5 mg capsules in amber glass bottles or in blister packs.
  Interventions: Drug: FK506E

INTERVENTIONS:
Drug: FK506E — oral
  Other Names: Astagraf XL; Advagraf; Graceptor; MR4; Prograf XL

SUMMARY:
The purpose of this study was to offer patients who had participated in one of the phase II PK or phase III studies on FK506E (MR4) the possibility to continue FK506E (MR4) until commercial availability of the drug and to record long term efficacy and safety data.

DETAILED DESCRIPTION:
The objective of this study was to asses the safety and efficacy of FK506E (MR4) as a long-term treatment in transplant recipients. Only patients who had participated in one of the phase II PK or phase III studies on FK506E (MR4) and had received at least one dose of study medication were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had already participated in the previous phase II pharmacokinetic or phase III studies with FK506E (MR4).
* Patients capable of understanding the purpose and risks of the study, who had been fully informed and given written informed consent to participate in the study.

Exclusion Criteria:

* Pregnant women or nursing mothers.
* Women unwilling or unable to use adequate contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2003-02-24 (Actual); Primary Completion 2009-10-07 (Actual); Study Completion 2009-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe Ltd.
Locations (102):
- University Hospital, Cincinnati, Ohio, United States
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Austria (2):
  - Landeskrankenhaus Innsbruck, Innsbruck
  - AKN Wien, Vienna
- Belgium (5):
  - Hospital Erasme, Brussels
  - Cliniques Universitaires St. Luc, Brussels
  - Departement Heelkunde, Ghent
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - Domaine Universitaire du Sart Tillman, Liège
- Brazil (4):
  - Hospital da Clínicas da UNICAMP, Campinas
  - Hospital São Francisco, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Geral de Bonsucesso, Rio de Janeiro
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Institut de Cardiologie de Montréal, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Vancouver Hospital & Health Sciences Centre, Vancouver
- IKEM, Prague, Czechia
- Skejby University Hospital, Århus N, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- France (16):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Bicetre Cedex
  - Hopital Saint-Eloi, Montpellier, Cedex 05
  - Hopital Laennec, Nantes, Cedex 1
  - Hotel Dieu, Nantes, Cedex 1
  - Service de Nephrologie, Nice, Cedex 1
  - Hôpital Edouard Hérriot, Lyon, Cedex 3
  - Hôpital Lapeyronie, Montpellier, Cedex 5
  - Hôpital Rangueil, Toulouse, Cedex 9
  - Hôpital Calmette, Lille, Cedex
  - Hopital Pontchaillou, Rennes, Cedex
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Chu Nord, Grenoble
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Hautepierre, Strasbourg
  - Hopital Paul Brousse, Villejuif
- Germany (15):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Universitätsklinik Charité, Berlin
  - Charite Campus Virchow Klinikum, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - DR MED Wolfgang Arns, Cologne
  - Medizinische Klink IV, Erlangen
  - Universitätklinikum Essen, Essen
  - Funktionsbereich Nephrologie, Frankfurt am Main
  - Univ. Klinik und Poliklinik fuer Urologie, Halle
  - Universitäts-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Leiter Viszerale Organtransplantation, Heidelberg
  - Klinikum Rechts der Isar, München
  - Klinik und Poliklinik fuer Chirurgie, Regensburg
  - Klinikum der Universität Regensburg, Regensburg
- Semmelweis University of Medicine, Budapest, Hungary
- Ireland (2):
  - National Liver Transplantation Unit, Dublin
  - Beaumont Private Clinic, Dublin
- Italy (10):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Unita Operativa Trapianto di Fegato e Multiorgano, Bologna
  - DISCAT - Centro Trapianti, Genova
  - Azienda Ospedaliera Ospedale Maggiore di Milano, Milan
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - Azienda Ospedaliera di Padova, Padua
  - ISMETT, Palermo
  - Policlinico Universitario Agostino Gemelli, Roma
  - Unita Operativa Complessa di Chirurgia dei Trapianti, Siena
  - Clinica Chirurgica Universitaria, Udine
- Mexico (2):
  - Instituto Mexicano de Transplantes Cuernava, Morelos
  - Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Tlalpan
- Akademisch Ziekenhuis Maastricht, Maastricht, Netherlands
- New Zealand Liver Transplant Unit, Auckland, New Zealand
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny, Szczecin
- South Africa (5):
  - Groote Schuur Hospital, Cape Town
  - Christiaan Barnard Memorial Hospital, Cape Town
  - St Augustine's Hospital, Durban
  - Jacaranda Hospital, Pretoria
  - University of Stellenbosch, Tygerberg Hospital, Tygerberg
- Spain (11):
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Servicio de Nefrologia, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Unidad de Trasplante Hepatico, Barcelona
  - Hospital General Universitario Gregorio Maranón, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Consultas de Trasplante Renal, Madrid
  - Hospital Central de Asturias, Oviedo
  - Clinica de Navarra, Pamplona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- Sweden (2):
  - SU/Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital Huddinge, Stockholm
- Universitätsspital Zürich, Zurich, Switzerland
- United Kingdom (7):
  - Walsgrove Hospital, Coventry
  - Queen Elizabeth Hospital, Edgbaston
  - Western Infirmary, Glasgow
  - Kings College Hospital, London
  - Department of Renal Medicine, Manchester
  - Wythenshaw Hospital, Manchester
  - The Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to Results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in 128 centers in 24 countries worldwide. The Principal Investigator at each study site was a medical doctor experienced in the treatment of transplant participants.
Pre-assignment Details: Only patients who had participated in one of the phase II PK or phase III studies on FK506E (MR4) and had received at least one dose of study medication were enrolled.
Groups:
- FG-506-11-01: Participants that had previously taken part in the FG-506-11-01 Phase II de novo liver transplant recipient study.
- FG-506E-12-01: Participants that had previously taken part in the FG-506E-12-01 Phase II de novo kidney transplant recipient study.
- FG-506E-12-02: Participants that had previously taken part in the FG-506E-12-02 Phase II kidney transplant recipient (Conversion from Prograf® to MR4) study.
- FG-506-15-02: Participants that had previously taken part in the FG-506-15-02 Phase II heart transplant recipient (Conversion from Prograf® to MR4) study.
- FG-506E-11-03: Participants that had previously taken part in the FG-506E-11-03 Phase III de novo liver transplant recipient study.
- FG-506E-12-03: Participants that had previously taken part in the FG-506E-12-03 Phase III de novo kidney transplant recipient study.
- PMR-EC-1105: Participants that had previously taken part in the PMR-EC-1105 Phase III liver transplant recipient (Conversion from Prograf® to MR4) study.
- PMR-EC-1205: Participants that had previously taken part in the PMR-EC-1205 Phase III kidney transplant recipient (Conversion from Prograf® to MR4) study.
- PMR-EC-1209: Participants that had previously taken part in the PMR-EC-1209 Phase III kidney transplant recipient (Conversion from cyclosporine A to MR4) study.
- PMR-EC-1210: Participants that had previously taken part in the PMR-EC-1210 Phase III de novo kidney transplant recipient study.
Period: Overall Study
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Started | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9
Completed | 30 | 32 | 53 | 55 | 113 | 163 | 83 | 105 | 84 | 7
Not Completed | 17 | 15 | 14 | 24 | 17 | 28 | 2 | 2 | 4 | 2
Not completed — Death | 4 | 0 | 4 | 6 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 4 | 5 | 5 | 9 | 1 | 1 | 4 | 0
Not completed — Consent withdrawn | 2 | 0 | 3 | 4 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 2 | 1 | 1 | 5 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Immunosuppressive regimen (not MR4) | 1 | 5 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 2
Not completed — Prohibited medication | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 1 | 2 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of the Full Analysis Set (FAS) population. The FAS included all subjects who received at least one dose of study drug, MR4, while participating in one of the phase II PK or phase III studies and at least one dose of MR4 during this study.
Groups:
- PMR-EC-1105: Participants that had previously taken part in the PMR-EC-1105 Phase III liver transplant recipient (Conversion from Prograf® to MR4) study. Participants that had previously taken part in the PMR-EC-1205 Phase III kidney transplant recipient (Conversion from Prograf® to
- Total: Total of all reporting groups
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210 | Total
Number analyzed (Participants) | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9 | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (9.5) | 44.0 (11.6) | 44.7 (12.4) | 51.3 (11.4) | 53.9 (8.4) | 46.9 (12.1) | 53.2 (10.3) | 49.4 (12.1) | 53.8 (11.1) | 36 (13.3) | 49.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 27 | 48 | 64 | 91 | 117 | 61 | 80 | 52 | 5 | 581
  Male | 11 | 20 | 19 | 15 | 39 | 74 | 24 | 27 | 36 | 4 | 269

OUTCOME MEASURES:

1. Primary Outcome: Participant Survival
Description: Participant survival was analyzed using Kaplan-Meier (KM) method procedures at 66 months (phase 2) and 24 months (phase III). The two-sided 95% confidence intervals (CI) for the estimated rates of patients alive at end of study (EOS) was calculated using Greenwood's formula. Start, event and censor times for the Kaplan-Meier analyses of participant survival were (Event time: day of death, Censor Time: day of last follow-up (for participants prematurely withdrawn from the study), and day of last visit (for participants completing the study) .
Time Frame: Up to 5.5 years (66 months (phase II) and 24 months (phase III)).
Population: The population for analysis was the Full Analysis Set (FAS) which included all subjects who received at least one dose of study drug, MR4, while participating in one of the phase II Pharmacokinetics (PK) or phase III studies and at least one dose of MR4 during this study.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Number analyzed (Participants) | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9
survival probability | 0.9092 [0.824 to 0.994] | 1.0000 [1.000 to 1.000] | 0.9356 [0.875 to 0.997] | 0.9031 [0.828 to 0.979] | 0.9536 [0.899 to 1.000] | 0.9933 [0.980 to 1.000] | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | NA [NA to NA] — No Kaplan-Meier estimates due to the short subject participation period and the low number of subjects.

2. Primary Outcome: Graft Survival
Description: Graft survival was analyzed using Kaplan-Meier Method procedures at 66 months (phase II) and 30 months (phase III). The two-sided 95% confidence intervals for the estimated rates of patients free from graft loss at EOS was calculated using Greenwood's formula. Graft loss was defined as re-transplantation or death. For kidney transplantation graft loss was also defined as nephrectomy or return to long-term dialysis. The date of graft loss is the earliest date of either of these events. Start, event and censor times for the Kaplan-Meier analyses of graft survival were (Event time: day of death, Censor Time: day of last follow-up (for participants prematurely withdrawn from the study), and day of last visit (for participants completing the study) .
Time Frame: Up to 5.5 years ((66 months (phase II) and 30 months (phase III)).
Population: Study analysis population for this primary endpoint consisted of the FAS.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Number analyzed (Participants) | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9
survival probability | 0.9092 [0.824 to 0.994] | 1.0000 [1.000 to 1.000] | 0.9217 [0.856 to .988] | 0.9031 [0.828 to 0.979] | 0.9536 [0.899 to 1.000] | 0.9469 [0.889 to 1.000] | 1.0000 [1.000 to 1.000] | 0.9898 [0.970 to 1.000] | 1.0000 [1.000 to 1.000] | NA [NA to NA] — No Kaplan-Meier estimates due to the short subject participation period and the low number of subjects.

3. Secondary Outcome: Biopsy-confirmed Acute Rejection (BCAR) Episodes
Description: FAS population. Evaluation of biopsy specimens performed by local histopathologist following "Histological Grading of Biopsies for Rejection" using grading relevant to type of organ allograft. Spontaneously resolving AR defined as episode not treated with new/increased corticosteroid medication, antibodies/any other medication and resolved irrespective of any MR4/MMF/azathioprine dose changes; corticosteroid sensitive AR was an episode which was treated with new/increased corticosteroid medication only and resolved, irrespective of any MR4, MMF or azathioprine dose changes; corticosteroid resistant AR was an episode which did not resolve following treatment with corticosteroids, if it was not treated with corticosteroids first but only with antibodies, it was included in this category; corticosteroid resistant AR episodes were further classified into episodes which resolved with further treatment and those which did not respond to further treatment/were ongoing at EOS/withdrawal.
Time Frame: Up to 6 years.
Population: FAS population.
Measure: Number; unit: participants with with BCAR episodes
Groups:
- PMR-EC-1210: Participants that had previously taken part in the PMR-EC-1210 Phase III de novo kidney transplant recipient study. There were no reported BCAR in subjects in the previous study PMR-EC-1210, Kaplan-Meier estimate not applicable.
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Number analyzed (Participants) | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9
participants with with BCAR episodes
  BCAR episodes | 3 | 3 | 0 | 9 | 5 | 1 | 0 | 0 | 1 | 0
  In male subjects N=36,27,48,64,91,117,61,80,52,5 | 2 | 1 | 0 | 9 | 3 | 0 | 0 | 0 | 1 | 0
  In female subjects N=11,20,19,15,39,74,24,27,36,4 | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  BCAR episodes with spontaneous resolution | 1 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0
  Corticosteriod sensitive BCAR episodes | 2 | 2 | 0 | 5 | 3 | 1 | 0 | 0 | 0 | 0
  Corticosteroid resistant BCAR episodes | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Mild histological grade of BCAR episodes | 2 | 1 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 0
  Moderate histological grade of BCAR episodes | 0 | 2 | 0 | 4 | 2 | 0 | 0 | 0 | 1 | 0
  Severe histological grade of BCAR episodes | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Unknown histological grade of BCAR episodes | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: FG-506-11-01; The two-sided 95% confidence interval for the estimated rate of freedom from BCAR at EOS was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method = 0.9257, 95% CI 2-sided [0.844 to 1.000]
Statistical Analysis 2: Comparison: FG-506E-12-01; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9321, 95% CI 2-sided [0.858 to 1.000]
Statistical Analysis 3: Comparison: FG-506E-12-02; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 1.0000, 95% CI 2-sided [1.0000 to 1.0000]
Statistical Analysis 4: Comparison: FG-506-15-02; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.8699, 95% CI 2-sided [0.790 to 0.949]
Statistical Analysis 5: Comparison: FG-506E-11-03; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9607, 95% CI 2-sided [0.927 to 0.995]
Statistical Analysis 6: Comparison: FG-506E-12-03; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9948, 95% CI 2-sided [0.985 to 1.000]
Statistical Analysis 7: Comparison: PMR-EC-1105; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 1.0000, 95% CI 2-sided [1.0000 to 1.0000]
Statistical Analysis 8: Comparison: PMR-EC-1205; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 1.0000, 95% CI 2-sided [1.0000 to 1.0000]
Statistical Analysis 9: Comparison: PMR-EC-1209; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9773, 95% CI 2-sided [0.933 to 1.000]

4. Secondary Outcome: Time to First BCAR Episode
Description: The time to first acute rejection episode was defined as the number of days from day 1 (defined as the day of study enrollment) to the first clinical, laboratory or histological signs that were considered to be related to the first acute rejection episode.
Time Frame: Up to 1344 days (3.75 years).
Population: The study analysis population for this endpoint consisted of subjects with biopsy confimed acute rejection.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Number analyzed (Participants) | 3 | 3 | 0 | 9 | 5 | 1 | 0 | 0 | 1 | 0
days | 479.3 (634.5) | 358 (350.8) |  | 601.2 (405.8) | 89.6 (148.4) | 1 (0) |  |  | 192 (0) |

5. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have a causal relationship with treatment. An AE was, therefore, any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use the study drug, whether or not related to the study drug. Causally-related is defined as a highly probably, probably, possible, not assessable or missing relationship as assessed by the investigator. An SAE was any untoward medical occurrence that at any dose: Resulted in death, was life threatening: did not refer to event which hypothetically might have caused death if more severe); resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect; required inpatient hospitalization/led to prolongation of hospitalization (treatment/observation/examination caused by AE was considered serious); other medically important events.
Time Frame: From first dose to duration of participation in the study (up to 6 years and 28 days after EOS).
Population: FAS population.
Measure: Number; unit: participants with adverse events
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Number analyzed (Participants) | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9
participants with adverse events
  Adverse events | 47 | 47 | 67 | 73 | 130 | 180 | 58 | 59 | 62 | 1
  Causally related adverse events | 47 | 42 | 44 | 56 | 112 | 132 | 33 | 29 | 21 | NA — No casually related AE summary data was available on subjects from previous study PMR-EC-1210 since the number of subjects was small and the study was still in progress at the time of the report.
  Serious adverse events | 36 | 31 | 40 | 43 | 67 | 64 | 13 | 16 | 15 | 2
  Causally related serious adverse events | 22 | 16 | 15 | 21 | 31 | 30 | 5 | 7 | 2 | NA — No casually related SAE summary data was available on subjects from previous study PMR-EC-1210 since the number of subjects was small and the study was still in progress at the time of the report.
  Deaths | 4 | 0 | 4 | 6 | 3 | 1 | 0 | 0 | 0 | 0

6. Post Hoc Outcome: Efficacy Failure
Description: Efficacy failure was defined as BCAR, graft loss, death, or an unknown outcome at the end of the study period. Start, event and censor times for the Kaplan-Meier analyses of efficacy failure were (Event time: onset of first episode of BCAR, graft loss, or death after study start, Censor Time: day of withdrawal (for participants prematurely withdrawn from the study), and day of last visit (for participants completing the study). No Kaplan-Meier estimates for PMR-EC-1210 due to the short subject participation period and the low number of subjects
Time Frame: Up to 5.75 years ((69 months (phase II) and 33 months (phase III)).
Population: The study analysis population for this endpoint consisted of participants with efficacy failure.
Measure: Number; unit: participants with efficacy failure
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Number analyzed (Participants) | 47 | 47 | 67 | 79 | 130 | 191 | 85 | 107 | 88 | 9
participants with efficacy failure
  Failure during the study | 6 | 3 | 5 | 15 | 8 | 6 | 0 | 1 | 1 | 0
  Failure after withdrawal | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Failure cause during study: BCAR | 3 | 3 | 0 | 9 | 5 | 2 | 0 | 0 | 1 | 0
  :Acute respiratory failure | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  :Astrocytoma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  :Chronic allograft dysfunction | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  :Hepatic cirrhosis | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  :Hypoglycemia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  :Increased creatinine | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  :Cerebrovascular accident | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  :Lymphoma | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  :Lung neoplasm | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  :Operative hemorrhage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  :Pulmonary embolism | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  :Renal insufficiency | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  :Sudden death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  :Cardiac disorder | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  :Hepatic insufficiency | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  :Hemolytic/uremic syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  :Esophageal varices hemorrhage | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  :Urethral stenosis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Failure cause after withdrawal: Lost to follow-up | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: FG-506-11-01; The two-sided 95% confidence interval for the estimated rate of freedom from efficacy failure at EOS was calculated using Greenwood's formula; Test type: Superiority or Other; Kaplan-Meier Method = 0.8391, 95% CI 2-sided [0.729 to 0.949]
Statistical Analysis 2: Comparison: FG-506E-12-01; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.8792, 95% CI 2-sided [0.778 to 0.981]
Statistical Analysis 3: Comparison: FG-506E-12-02; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.8816, 95% CI 2-sided [0.782 to 0.981]
Statistical Analysis 4: Comparison: FG-506-15-02; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.7769, 95% CI 2-sided [0.675 to 0.878]
Statistical Analysis 5: Comparison: FG-506E-11-03; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.8373, 95% CI 2-sided [0.693 to 0.981]
Statistical Analysis 6: Comparison: FG-506E-12-03; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9419, 95% CI 2-sided [0.883 to 1.000]
Statistical Analysis 7: Comparison: PMR-EC-1105; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 1.0000, 95% CI 2-sided [1.000 to 1.000]
Statistical Analysis 8: Comparison: PMR-EC-1205; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9898, 95% CI 2-sided [0.970 to 1.000]
Statistical Analysis 9: Comparison: PMR-EC-1209; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Kaplan-Meier Method = 0.9773, 95% CI 2-sided [0.933 to 1.000]

ADVERSE EVENTS:
Time Frame: From first dose to duration of participation in the study (up to 6 years and 28 days after EOS).
Description: FAS population, Treatment Emergent Events only. The following adverse events (AEs) are excluded from summary: 'Kidney transplant rejection', 'Heart transplant rejection', 'Liver transplant rejection', and 'Transplant rejection'.
Arm/Group | FG-506-11-01 | FG-506E-12-01 | FG-506E-12-02 | FG-506-15-02 | FG-506E-11-03 | FG-506E-12-03 | PMR-EC-1105 | PMR-EC-1205 | PMR-EC-1209 | PMR-EC-1210
Serious Adverse Events (participants affected / at risk) | 36/47 | 31/47 | 40/67 | 43/79 | 67/130 | 64/191 | 13/85 | 16/107 | 15/88 | 2/9
Other Adverse Events (participants affected / at risk) | 47/47 | 47/47 | 66/67 | 73/79 | 129/130 | 175/191 | 52/85 | 54/107 | 60/88 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FG-506-11-01 (N=47) | FG-506E-12-01 (N=47) | FG-506E-12-02 (N=67) | FG-506-15-02 (N=79) | FG-506E-11-03 (N=130) | FG-506E-12-03 (N=191) | PMR-EC-1105 (N=85) | PMR-EC-1205 (N=107) | PMR-EC-1209 (N=88) | PMR-EC-1210 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Bone marrow depression (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Secondary anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery atherosclerosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vestibular neuronitis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Internal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 6 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic artery occlusion (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic artery stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic oedema (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Bakulovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Bronchitis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 4 | 0 | 0 | 3 | 1 | 0 | 2 | 0
Gastroenteritis Norwalk virus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoid infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 3 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Histoplasmosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human polyomavirus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected lymphocele (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective thrombosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotid abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis carinii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 1 | 3 | 1 | 4 | 0 | 1 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shunt infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 9 | 2 | 0 | 0 | 7 | 0 | 1 | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye penetration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 3 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose fluctuation (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis acquired (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
B-cell unclassifiable lymphoma high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain mass (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 2 | 1 | 0
Renal insufficiency (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Renal vessel disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vesico-ureteric reflux (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Emphysematous bulla (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol detoxification (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cataract extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreas transplant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Iliac artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leriche syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebothrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FG-506-11-01 (N=47) | FG-506E-12-01 (N=47) | FG-506E-12-02 (N=67) | FG-506-15-02 (N=79) | FG-506E-11-03 (N=130) | FG-506E-12-03 (N=191) | PMR-EC-1105 (N=85) | PMR-EC-1205 (N=107) | PMR-EC-1209 (N=88) | PMR-EC-1210 (N=9)
Anaemia (Blood and lymphatic system disorders) | 11 | 9 | 5 | 9 | 11 | 21 | 0 | 5 | 4 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 14 | 5 | 0 | 1 | 11 | 5 | 0 | 0 | 0 | 1
Secondary anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 4 | 9 | 3 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 5 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 4 | 1 | 5 | 0 | 0 | 0 | 0
Melanocytic naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 2 | 3 | 7 | 4 | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 0 | 5 | 1 | 5 | 3 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 7 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 2 | 4 | 4 | 4 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 8 | 5 | 23 | 12 | 24 | 2 | 3 | 12 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 5 | 5 | 2 | 6 | 2 | 1 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 1 | 4 | 17 | 8 | 2 | 1 | 1 | 0 | 0
Oral soft tissue disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pancreas lipomatosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 3 | 11 | 2 | 6 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 1 | 8 | 4 | 3 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 9 | 8 | 7 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 4 | 11 | 7 | 15 | 8 | 19 | 1 | 2 | 4 | 1
Pyrexia (General disorders) | 6 | 3 | 2 | 6 | 6 | 6 | 0 | 3 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 6 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 5 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 1 | 6 | 2 | 7 | 2 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 4 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 4 | 1 | 1 | 1 | 6 | 1 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0
Hepatitis C (Infections and infestations) | 8 | 0 | 0 | 0 | 22 | 2 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 4 | 2 | 1 | 1 | 2 | 7 | 1 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 4 | 12 | 8 | 5 | 6 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 16 | 3 | 15 | 7 | 12 | 0 | 1 | 4 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 4 | 2 | 4 | 1 | 6 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 7 | 1 | 3 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 5 | 7 | 3 | 1 | 0 | 0 | 2 | 0
Skin bacterial infection (Infections and infestations) | 4 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 4 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 4 | 3 | 1 | 5 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 4 | 19 | 10 | 3 | 4 | 28 | 2 | 2 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 6 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 3 | 9 | 1 | 5 | 13 | 21 | 0 | 4 | 3 | 0
Blood glucose increased (Investigations) | 0 | 2 | 1 | 4 | 1 | 1 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 8 | 3 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 3 | 2 | 2 | 4 | 6 | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 0 | 2 | 4 | 7 | 2 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 4 | 5 | 4 | 3 | 9 | 4 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 4 | 4 | 8 | 1 | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 6 | 0 | 0 | 1 | 1
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 10 | 3 | 1 | 3 | 14 | 8 | 0 | 0 | 0 | 0
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 6 | 5 | 5 | 6 | 14 | 12 | 3 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 3 | 6 | 0 | 3 | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1
Gout (Metabolism and nutrition disorders) | 1 | 3 | 12 | 11 | 2 | 5 | 2 | 1 | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 9 | 11 | 0 | 4 | 14 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 12 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 5 | 0 | 2 | 7 | 17 | 3 | 2 | 1 | 0
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 2 | 2 | 1 | 6 | 2 | 3 | 2 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 6 | 4 | 3 | 9 | 18 | 2 | 4 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 13 | 1 | 0 | 12 | 13 | 8 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 5 | 1 | 5 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 4 | 4 | 1 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3 | 12 | 7 | 11 | 1 | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 3 | 20 | 14 | 7 | 1 | 2 | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 4 | 3 | 2 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 10 | 2 | 1 | 1 | 0 | 3 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 1 | 0 | 8 | 6 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 10 | 4 | 6 | 0 | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 5 | 1 | 2 | 0 | 2 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 15 | 2 | 3 | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 11 | 4 | 1 | 12 | 12 | 8 | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Nervous system disorders) | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 11 | 13 | 1 | 3 | 8 | 13 | 1 | 0 | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 8 | 2 | 10 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 4 | 4 | 4 | 13 | 5 | 3 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 2 | 6 | 6 | 8 | 5 | 2 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0 | 2 | 8 | 1 | 1 | 2 | 2 | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 4 | 1 | 1 | 2 | 5 | 0 | 5 | 3 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 4 | 3 | 0 | 6 | 6 | 5 | 2 | 0 | 2 | 0
Renal insufficiency (Renal and urinary disorders) | 12 | 1 | 0 | 7 | 25 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 1 | 12 | 6 | 7 | 2 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 10 | 2 | 2 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 0 | 3 | 5 | 0 | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 8 | 5 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 7 | 1 | 2 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 4 | 1 | 3 | 0 | 0 | 0 | 0
Nasal sinus drainage (Surgical and medical procedures) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 19 | 11 | 13 | 19 | 50 | 41 | 13 | 6 | 4 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 4 | 2 | 3 | 0 | 2 | 0 | 0
Secondary hypertension (Vascular disorders) | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 0 | 0 | 6 | 0 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
No Kaplan-Meier estimates for PMR-EC-1210 due to the short subject participation period and the low number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained during the conduct of the study is regarded as confidential. Agreement from the sponsor is required prior to disclosing any information relevant to the study.